CLINICAL TRIAL: NCT05499104
Title: A Prospective, Randomized, Controlled Trial Comparing a Cellulose Dressing to Two Standard of Care Dressings in Treating Split Thickness Donor Sites in Burn and Wound Patients.
Brief Title: A Trial Comparing a Cellulose Dressing to Two Standard of Care Dressings in Treating Split Thickness Donor Sites in Burn and Wound Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joseph M. Still Research Foundation, Inc. (Other)
Collaborators: Innovatech Engineering, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMSRF-NCMIS-P01
Record Dates: First submitted 2021-07-20; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Donor Sites; Wound Heal; Wound Drainage; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Mepilex Ag (Active Comparator): patient will receive Mepilex Ag for their site, standard of care to be followed.
  Interventions: Device: Mepilex Ag
- Xeroform (Active Comparator): patient will receive Xeroform for their site, standard of care to be followed.
  Interventions: Device: Xeroform
- NovaDress (Experimental): patient will receive NovaDress for their site, standard of care to be followed.
  Interventions: Device: NovaDress

INTERVENTIONS:
Device: NovaDress — NovaDress is constructed of pure cellulose derived from tree pulp. The tree pulp is reconstructed into hydrated sheets wrapped in nonwoven viscose and irradiated.
  Arms: NovaDress
Device: Mepilex Ag — Mepilex Ag is an antimicrobial foam dressing that absorbs low to moderate exudate and maintains a moist wound environment.
  Arms: Mepilex Ag
Device: Xeroform — Xeroform® Occlusive Dressing (XF) is a fine-mesh gauze impregnated with a petrolatum blend, 3% bismuth tribromophenate.
  Arms: Xeroform

SUMMARY:
This is a three arm study, comparing the Novadress, Mepilex Ag, and Xeroform Occlusive dressings for healing, drainage, and pain management. NovaDress is constructed of pure cellulose derived from tree pulp. Mepilex Ag is a antimicrobial foam dressing that absorbs low to moderate exudate and maintains a moist wound environment. Xeroform Occlusive Dressing is a fine-mesh gauze impregnated with a petrolatum blend, 3% bismuth tribromophenate.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years of age.
* Has been admitted to the Joseph M. Still Burn Center at Doctors Hospital Augusta or The Advanced Wound Clinic, needing a split-thickness skin graft and will undergo a subsequent donor site harvest.
* Subject is able to provide informed consent.
* Has a negative urine or serum pregnancy test at screening (if female and has potential for pregnancy) if available or if stated by patient.

Exclusion Criteria:

* Has a Baux Score of ≥130.
* Subject is intubated, unable to state pain levels.
* Has active diagnosis of any autoimmune process, cancer, or organ failure that in the opinion of the investigator would prevent the subject from successfully participating in the study,
* Has coagulopathy that in the opinion of the investigator, would place subject at an increased risk for bleeding.
* Vulnerable subjects who, in the opinion of the Investigator, present with poor skin integrity (i.e. Elderly), is a prisoner, non-English speaking, or is without means of follow-up or return to clinic (i.e. homeless).
* Is pregnant, plans to become pregnant, or is actively breastfeeding.
* Active illicit drug use.
* Is moribund, or in the opinion of the investigator is not expected to survive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Pain and Healing | 14 days
  To compare and healing (defined as >95% epithelization) at the study donor sites treated with a cellulose dressing to two standard of care dressings- an antimicrobial foam dressing and a bacteriostatic petrolatum based gauze dressing.

SECONDARY OUTCOMES:
Absorbent ability | 14 days
  Ability of dressing to absorb exudate measured by staff satisfaction survey
Conformability | 14 days
  Ability of dressing to maintain shape measured by staff satisfaction survey
Adherence | 14 days
  Ability of dressing to remain fixed in place measured by staff satisfaction survey
Management of bloody exudate | 14 days
  Ability of dressing to absorb bloody exudate measured by staff satisfaction survey
Ease of removal | 14 days
  Ability of dressing to be removed in an atraumatic fashion measured by staff satisfaction survey
Cost | 14 days
  Average cost incurred by the patient for donor site dressings measured by staff satisfaction survey

CONTACTS AND LOCATIONS:
Locations (1):
- Joseph M. Still Research Foundation, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No